CLINICAL TRIAL: NCT03670407
Title: Follicular Activation by Fragmentation of Ovarian Tissue
Acronym: FAFOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Podobnik Maternity and Gynecology Hospital (Other)
Responsible Party: Principal Investigator, Miro Šimun Alebić, Head of human reproduction unit, Podobnik Maternity and Gynecology Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201810001
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Diminished Ovarian Reserve
Keywords: Premature Ovarian Failure; Infertility, Female; Ovarian tissue fragmentation
MeSH Terms: conditions — Primary Ovarian Insufficiency; Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants who opt not to go ahead with ovarian fragmentation.
- Study group (Experimental): Participants who opt for ovarian fragmentation.
  Interventions: Procedure: Ovarian tissue fragmentation

INTERVENTIONS:
Procedure: Ovarian tissue fragmentation — Unilateral ovariectomy, ovarian tissue in vitro fragmentation and reimplantation.
  Arms: Study group

SUMMARY:
The primary objective of this study is to assess the chances of increasing the number of antral follicles in ovarian tissue of patients with diminished ovarian reserve by activation of primordial follicles through ovarian cortex fragmentation. Secondary objectives are to assess potential association with the number of oocytes retrieved and pregnancy rates after IVF.

ELIGIBILITY:
Inclusion Criteria:

1. previous ≥ 2 poor ovarian responds (≤ 3 retrieved oocytes) in an antagonist cycle with a minimum of 225 IU gonadotropins a day or corifollitropin 150 mcg) in patients >35 i <40 years
2. previous cycle with ≤ 3 retrieved oocytes) in an antagonist cycle with a minimum of 225 IU gonadotropins a day or corifollitropin 150 mcg) in patients >35 i <40 years with antral follicle count (AFC) ≤ 5 i/ili antiM¸ulelrian hormone (AMH) ≤ 6.5pmol/L
3. premature ovarian insufficiency according to European Society of Human Reproduction and Embryology (ESHRE) development group, 2015 in patients 18-40 years
4. undetectable AMH serum levels and follitropin (FSH) >35 IU/ml in two serum samples separated by at least 4 weeks

Exclusion Criteria:

1. clinical/ultrasonographical signs of endometriosis
2. previous ovarian/pelvic surgery
3. previous gonadotoxic treatment
4. genito-urinary tract malformations
5. extreme male infertility ( <10 000 progressively motile sperms in the semen sample)
6. inform consent unsigned -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Antral follicle count | 6 months

SECONDARY OUTCOMES:
The number of oocytes retrieved | 1 year
Clinical pregnancy rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Miro S Alebić, Principal Investigator — Podobnik Maternity and Gynecology Hospital
Locations (1):
- Podobnik Maternity and Gynecology Hospital, Zagreb, Croatia